CLINICAL TRIAL: NCT07268183
Title: Influence of Pre-diagnostic Estrogen Fluctuations on the Development of Prolactin-Secreting Macroadenomas or Microadenomas: A Comparative Study Conducted at Hôpital Louis Pradel
Brief Title: How Estrogen Fluctuations Before Diagnosis Affect the Size Prolactin-secreting Tumors
Acronym: OEMacroPrL
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0853
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Prolactinoma; Macroprolactinoma
Keywords: Prolactinoma; Macroprolactinoma; pituitary adenomas; lactotroph adenoma; risk factor; microprolactinoma; Combined hormonal contraception; combined oral contraception; estrogen impact
MeSH Terms: conditions — Prolactinoma; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with a macroprolactinoma: Women with prolactin-producing macroadenomas diagnosed between 2013 and 2023 Followed by the Hospices Civiles de Lyon, Hôpital Cardiologique of Bron.
  Interventions: Other: Standardized questionnaire
- Women with a microprolactinoma: Women with prolactin-producing microadenomas diagnosed between 2013 and 2023 Followed by the Hospices Civiles de Lyon, Hôpital Cardiologique of Bron.
  Interventions: Other: Standardized questionnaire

INTERVENTIONS:
Other: Standardized questionnaire — The intervention is a questionnaire which will be administered only if informations available on medical files are not sufficient.
  1 mounth before questionning our cases and controls, they will receive a participant information note.
  It will be administered primarily by telephone. If the patient prefers not to answer by telephone, a paper version will be mailed to her. In this case, she will have up to two months to return the completed questionnaire by post.
  The questionnaire will collect detailed information on potential exposures to estrogens and reproductive history.

SUMMARY:
Prolactinomas are the most common pituitary adenomas, representing about two-thirds of clinically relevant cases. Their prevalence is around 50 per 100,000 individuals, with an incidence of 3-5 new cases per 100,000 per year and has been rising in recent decades.

They may increase morbidity and mortality due to several factors:

* Hormone hypersecretion: excess prolactin causes galactorrhea, amenorrhea, and infertility.
* Mass effect: macroadenomas can compress adjacent structures, leading to headaches, visual loss, or neurological symptoms.
* Treatment complications: medical or surgical treatments may carry risks.

A marked sex difference exists, with a male-to-female ratio of 1:5-1:10, and peak diagnosis in women aged 25-44. This disparity disappears after menopause, supporting a potential role of estrogens in tumor development. Lactotrope cells, from which prolactinomas arise, are estrogen-sensitive, unlike other pituitary tumor cells (e.g., somatotrophs, gonadotrophs).

A large 2022 prospective cohort (nurses) suggested a possible association between pituitary adenomas and both combined oral contraceptives (COCs) and hormone therapy (HT). However, limitations included self-reported diagnoses, lack of adenoma characterization, and contradictory findings (association with HT but not consistently with COCs). A 2009 case-control study including all adenomas found no link with hormonal contraception, while older studies from the 1980s assessed high-dose contraceptives no longer in use.

Microprolactinomas are 4-5 times more frequent than macroprolactinomas (≥10 mm). Distinguishing between the two is essential, as they differ in clinical presentation, prognosis, and sex distribution. Macroadenomas are more common in men, possibly due to delayed diagnosis, as symptoms such as decreased libido are less specific, whereas women often present with amenorrhea or galactorrhea. However, studies suggest tumor size is not directly linked to symptom duration, indicating other factors may explain macroadenoma development.

Why some patients develop macro- rather than microadenomas remains unclear. Estrogen exposure is a possible explanation. It is therefore relevant to investigate whether women with macroprolactinomas had greater exposure to endogenous estrogens (early menarche, late menopause, pregnancies, breastfeeding) or exogenous estrogens (contraception, menopausal HT) compared to women with microprolactinomas.

The hypothesis is that women with macroprolactinomas were exposed to higher cumulative levels of estrogens before diagnosis than women with microprolactinomas.

ELIGIBILITY:
Inclusion Criteria of cases :

* Female patients aged ≥ 18 years at recruitment (diagnosis may have occurred before age 18).
* Diagnosis of a prolactin-secreting macroadenoma established between January 2013 and December 2023. The diagnosis may have been made either in the Endocrinology Department of Hôpital Louis Pradel or by another medical team, whether within or outside the hospital setting. However, follow-up or part of the follow-up must have been performed in the Endocrinology Department of Hospices Civils de Lyon (HCL)
* Diagnosis established by : A hypothalamic-pituitary MRI centered on the sella turcica, performed with gadolinium injection, including fine T1-weighted coronal and sagittal slices (1.5-3 mm), showing an adenoma with at least one axis measuring > 10 mm, AND Serum prolactin > 100 µg/L, or 24-100 µg/L with either a favorable response to medical therapy or histopathological confirmation after surgery.
* Ability to understand the study and provide informed non-opposition.

Inclusion Criteria of controls :

* Female patients aged ≥ 18 years at the time of recruitment (diagnosis may have occurred before age 18).
* Diagnosis of a prolactin-secreting microadenoma established between January 2013 and December 2023. The diagnosis may have been made in any medical center, but follow-up or part of the follow-up must have been carried out in the Endocrinology Department of Hôpital Louis Pradel.
* Diagnosis must be based on: A hypothalamic-pituitary MRI centered on the sella turcica, performed with gadolinium injection, including fine T1-weighted coronal and sagittal slices (1.5-3 mm), showing a prolactin-secreting adenoma with all axes measuring < 10 mm, AND A biological assessment performed outside any condition likely to bias results (significant stress, physical exertion, pregnancy, or intake of hyperprolactinemia-inducing drugs unrelated to prolactinoma treatment), showing serum prolactin > 24 µg/L.
* Ability to understand the nature and implications of the study and to provide informed non-opposition to participation.

Exclusion Criteria of cases :

* Presence of a non-secreting macroadenoma.
* History of isolated hyperprolactinemia or an isolated pituitary lesion documented prior to 2013, without subsequent direct diagnosis of prolactinoma.
* Presence of a known genetic abnormality or a genetic syndrome predisposing to the development of a prolactin-secreting adenoma.

Exclusion Criteria of controls :

* Presence of a non-secreting microadenoma.
* Uncertain diagnosis of adenoma with an ongoing therapeutic trial.
* Isolated hyperprolactinemia without evidence of adenoma.
* Hyperprolactinemia or pituitary lesion without hyperprolactinemia documented prior to 2013, without subsequent direct diagnosis of prolactinoma.
* Presence of a known genetic abnormality or a genetic syndrome predisposing to the development of a prolactin-secreting adenoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in this study will be identified from the COLLEMARA database, used within the Hospices Civils de Lyon. This database, specifically dedicated to rare diseases, provides a structured registry of patients followed for rare pituitary disorders, such as prolactinomas.
  For the purpose of this study, the COLLEMARA database will be used solely to identify eligible patients, based on the coded diagnosis of "prolactinoma." The study population will consist of female patients whose diagnosis was made between 2013 and 2023 and who meet the other inclusion criteria.
  A total of 180 patients will be included: 60 in the case group ("macroprolactinomas") and 120 in the control group ("microprolactinomas").
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
number of patients exposed to combined estrogen-progestin contraception | week 4
  Identify the estrogen-dependent risk factor
number of patients exposed to menopausal hormone therapy | week 4
  Identify the estrogen-dependent risk factor
number of patients exposed to progestin-only treatment | week 4
  Identify the estrogen-dependent risk factor
number of patients exposed to Ovarian Stimulation | week 4
  Identify the estrogen-dependent risk factor
Age at First Use of Hormonal Contraception | week 4
  Identify the estrogen-dependent risk factor
Age at Menarche | week 4
  Identify the estrogen-dependent risk factor
Age at Menopause | week 4
  Identify the estrogen-dependent risk factor
Age at First Live Birth | week 4
  Identify the estrogen-dependent risk factor
Nulliparity | week 4
  Identify the estrogen-dependent risk factor
Number of Pregnancies Carried to Viability | week 4
  Identify the estrogen-dependent risk factor
Exposure to Breastfeeding defined as the total cumulative duration of breastfeeding across all pregnancies, expressed in months. • None: 0-1 month • Moderate: 1-12 months • High: >12 months | week 4
  Identify the estrogen-dependent risk factor

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Louis Pradel, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No